CLINICAL TRIAL: NCT01265485
Title: An Open Label Study to Examine the Effect of Coated Suppositories on Anal Pressure in Healthy Subjects
Brief Title: An Study to Examine the Effect of Coated Suppositories on Anal Pressure in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RDD Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDD 107
Record Dates: First submitted 2010-12-07; First posted 2010-12-23 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental)
  Interventions: Drug: coated suppository

INTERVENTIONS:
Drug: coated suppository — Dose escalating study

SUMMARY:
This is an open label, dose-finding, 2-parts study. Approximately 6 subjects will be participating in this study. This study is composed of 2 parts:

Part 1 is a dose finding study. Part 2 is a pharmacodynamic and pharmacokinetic study of an elected dose. A screening will be used to determine patients' suitability for inclusion in the trial. Within one week after the screening visit, subjects who meet all inclusion criteria and none of the exclusion criteria will enter part 1 of the study, one day of dose escalation. During this part, patients will undergo rectal manometry to determine anal pressure at baseline. Afterwards coated suppositories at various drug concentrations will be inserted and follow up manometries will be performed to determine response.

Patients that presented with an increase in rectal resting pressure without adverse events will enter the second part of the study. In this part, patients will be administered with a coated suppository, at a dose found at part 1 of the study to cause significant anal contraction. Manometry studies will be performed before insertion (baseline) and at 1, 3 and 5 hours after insertion.

Blood levels for drug concentrations will be taken at times 0, 30, 60, 120, 180, 300 minutes after administration and rectal manometries will be done at times 0, 1, 3 and 5 hours after administration.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Male or female subjects 18 to 55 years of age;

Exclusion Criteria:

* Known allergy to the active drug or excipients.
* Pregnancy or lactation.
* Active cardiovascular or cerebrovascular disease including unstable angina, myocardial infarction, transient ischemic attacks/stroke, clinically significant arrhythmia, congestive heart failure, or cardiac valve abnormalities;
* Type 1 diabetes mellitus;
* Insulin treated type 2 diabetes mellitus;
* Renal insufficiency.
* Liver insufficiency.
* Malignant disease within 5 years of screening;
* History of rectal surgery.
* History of HIV, hepatitis B, hepatitis C.
* Has upon physical examination a rectal deformation or signs of rectal disease such as fissure, bleeding hemorrhoids, fistula, infection or space occupying lesion.
* Chronic use of medications with the exception of birth control pills.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in resting anal pressure | 1 day
  The primary outcome is the change in resting anal pressure as measured 90 minutes after insertion of coated suppository and in comparison to baseline measurement taken before intervention.

SECONDARY OUTCOMES:
Drug absorption | 1 day
  Blood samples for determining drug absorption be taken at times 0, 30, 60, 120, 180, 300 minutes after administration

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shapiro, MD, Principal Investigator — Gastroenetrology dept, Asaf Harofe Medical Center
Locations (1):
- Gastroeneterology dept, Asaf harofe Medical center, Zrifin, Israel